CLINICAL TRIAL: NCT04167098
Title: A Prospective Randomized Placebo-controlled Trial Comparing Platelet-rich Plasma and Corticosteroid Injection for Treatment of Trigger Finger
Brief Title: Effectiveness of Platelet-rich Plasma for Treatment of Trigger Finger
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Töölö Hospital (Other)
Responsible Party: Principal Investigator, Samuli Aspinen, Principal investigator, Töölö Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2845/2019
Record Dates: First submitted 2019-11-10; First posted 2019-11-18 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Tendon Entrapment
Keywords: Platelet-Rich Plasma; Trigger Finger
MeSH Terms: conditions — Tendon Entrapment; Trigger Finger Disorder | interventions — Adrenal Cortex Hormones

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Platelet-Rich Plasma (Experimental)
  Interventions: Other: PRP injection
- Corticosteroid (Active Comparator)
  Interventions: Other: Corticosteroid injection
- 0.9% saline (Placebo Comparator)
  Interventions: Other: Placebo injection

INTERVENTIONS:
Other: PRP injection — 0.5 ml Platelet-rich Plasma around A1 tendon sheath
  Arms: Platelet-Rich Plasma
Other: Corticosteroid injection — 0.5 ml methylprednisolone around A1 tendon sheath
  Arms: Corticosteroid
Other: Placebo injection — 0.5 ml 0.9% saline around A1 tendon sheath
  Arms: 0.9% saline

SUMMARY:
Study purpose is to evaluate the effectiveness of Platelet-rich Plasma (PRP) injection in the treatment of trigger finger. We compare PRP to a corticosteroid (methylprednisolone) injection in a prospective randomized triple-blind placebo-controlled study.

Patients with clinically confirmed trigger finger are randomized (1:1:1 computer generated sequence with random block size) to three parallel groups and will receive an injection of either PRP, corticosteroid or placebo (0.9% saline) around the affected tendon sheath in a double-blind setting.

Baseline data is collected and is followed by a phone call at 1 month, and follow-up visits at 3, 6, 12 and 24 months after the intervention. Unveiling of the allocation is at 6 months post-intervention.

The primary outcome measures are:

* Symptom resolution
* Patient-Rated Wrist Evaluation

Secondary outcomes:

* Quick-Disabilities of the Arm, Shoulder and Hand
* Pain Visual Analogue Score
* Global improvement (7-step Likert-scale)
* Grip strength
* Finger range of motion

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 75
* Symptom duration > 3 months

Exclusion Criteria:

* Diabetes
* Rheumatoid arthritis or other condition requiring continuous oral corticosteroids
* Previous history of surgery or injection to the affected ray
* Alcohol or drug abuse
* Mental instability

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Estimated)
Dates: Start 2019-11-01 (Actual); Primary Completion 2021-07-01 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
Symptom resolution | 24 months
  4-step Likert (0 = no response; 1 = partial response, but not satisfactory, warranting further treatment; 2 = partial response, satisfactory, not warranting further treatment; 3 = complete resolution of symptoms and signs)
Patient-Rated Wrist Evaluation | 24 months
  The PRWE comprises 15 questions to measure wrist pain and disability in daily activities. In PRWE patients rate wrist pain and disability from 0 to 10 and it consists two subscales: Pain and Function (0=best possible outcome, 10=worst possible outcome)

SECONDARY OUTCOMES:
Quick-Disabilities of the Arm, Shoulder and Hand | 24 months
  he QuickDASH is self-reported questionnaire and shortened version of DASH outcome measure to measure physical function and symptoms in people with any or multiple musculoskeletal disorders of the upper limb in 11 dimensions in 1-5 scale (1=best possible outcome, 5=worst possible outcome)
Pain (Visual Analogue Scale) | 24 months
  The VAS is derived by health care professional question of pain in scale 0 to 10 (0=no pain, 10=worst possible pain).
Global improvement | 24 months
  Global rating to treatment effect will be evaluated by question: "How would you rate the function of your hand compared to the situation before the treatment?". The options are in 5-step Likert scale from (-2) Much worse to (+2) Much better
Grip strength | 24 months
  Grip strength is measured with a dynamometer in kg as the mean of three measurements. It will be numbered in kg and percentage of the unaffected side.
Finger range of motion (ROM) | 24 months
  The ROM of the finger is measured on both hands with a handheld goniometer in degrees.

CONTACTS AND LOCATIONS:
Locations (1):
- Töölö Hospital (Helsinki University Hospital), Helsinki, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Aspinen S, Nordback PH, Anttila T, Stjernberg-Salmela S, Ryhanen J, Kosola J. Platelet-rich plasma versus corticosteroid injection for treatment of trigger finger: study protocol for a prospective randomized triple-blind placebo-controlled trial. Trials. 2020 Nov 27;21(1):984. doi: 10.1186/s13063-020-04907-w. PMID 33246497